CLINICAL TRIAL: NCT04073095
Title: Comparison of Ultrasound-Guided Modified-Thoracolumbar Interfascial Plane Block And Lumbar Erector Spinae Plane Block for Pain Management Following Lumbar Spinal Surgery
Brief Title: Erector Spinae Plane Block and Modified-Thoracolumbar Interfascial Plane Block Following Lumbar Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 2
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar spinal surgery; Postoperative pain management; Erector spina plane block; Modified thoracolumbar interfacial plane block
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: There are three models for this study. The first group is erector spinae plane block group, the second one is modified-thoracolumbar interfascial plane block, the third group is the no intervention control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group T = mTLIP block group (Active Comparator): In group T, mTLIP block will be performed. US probe will be placed vertically at the L3 vertebrae level. After visualizing the hyperechoic shadow of the spinous process and interspinous muscles as an anatomical guide point, the probe will be moved forward to the lateral to visualize the longissimus and iliocostal muscles. Between these muscles, block needle will be inserted within in plane technique in a medial-to-lateral direction in the interfascial plane. Once the needle tip will be placed within the interfacial plane and after careful aspiration to rule out intravascular needle placement, 2 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 20 mL will be injected in each side (total 40 mL).
  Interventions: Other: modified-thoracolumbar interfascial plane block (Group T)
- Group E = ESPB group (Active Comparator): In group E, ESP block will be performed. US probe will be placed longitudinally 2-3 cm lateral to the L3 transverse process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle will be inserted cranio caudal direction and then for correction of the needle 2 ml saline will be enjected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 20 ml %0.25 bupivacaine will be administered for block in each side (total 40 mL).
  Interventions: Other: Erector spinae plane block (Group E)
- Group C = Control group (No Intervention): Patients in control group will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period.A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.

INTERVENTIONS:
Other: Erector spinae plane block (Group E) — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period.A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 1, 2, 4, 8, 16 and 24 hours. If the VAS score will be ≥ 4, 0.5 mg/ kg meperidine IV will be administered. The first time of the use of rescue analgesic, intraoperative and postoperative opioid consumption, side effects such as nausea, vomiting, itching and block related complications will be recorded.
  Arms: Group E = ESPB group
Other: modified-thoracolumbar interfascial plane block (Group T) — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period.A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 1, 2, 4, 8, 16 and 24 hours. If the VAS score will be ≥ 4, 0.5 mg/ kg meperidine IV will be administered. The first time of the use of rescue analgesic, intraoperative and postoperative opioid consumption, side effects such as nausea, vomiting, itching and block related complications will be recorded.
  Arms: Group T = mTLIP block group

SUMMARY:
Ultrasound (US)-guided peripheral nerve blocks have been used increasily due to the advantages of ultrasound in anesthesia practice. TLIP block is one of these nerve blocks performed under US guidance. In this technique, local anesthetic solution is injected between the multifidus and logissimus muscles nearly at the level of the 3rd lumbar vertebra and targets the dorsal rami of the thoracolumbar nerves. However, the visualisation of this technique may be difficult under US guidance. Therefore, modified-TLIP (mTLIP) block was defined as a new approach. It has been reported that mTLIP block may provide effective analgesia management after lumbar spine surgery.

The ultrasound (US) guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. at 2016. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. It has been reported that ESPB provides lumbar analgesia at T10-12, L3. The aim of this study is to compare US-guided mTLIP block and ESPB pain management after lumbar discectomy+ surgery.

DETAILED DESCRIPTION:
Spine surgery in thoracolumbar region is one of the most common surgeries performed for the treatment of leg and back pain. Pain management is especially important for these patients since chronic pain often occurs after surgery. Severe pain may occur at postoperative period in patients following lumbar disc herniation (LDH) operation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Opioids are one of the most preferred drugs among the analgesic agents. Parenteral opioids are generally performed for patients after surgery. However opioids have undesirable adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events).

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment. US-guided interfascial plane blocks have been used increasily due to the advantages of ultrasound in anesthesia practice. TLIP block is one of these nerve blocks performed under US guidance and defined by Hand et al. in 2015. In this technique, local anesthetic solution is injected between the multifidus and logissimus muscles nearly at the level of the 3rd lumbar vertebra and targets the dorsal rami of the thoracolumbar nerves. However, the visualisation of this technique may be difficult under ultrasound (US) guidance. Therefore, Ahiskalioglu et al. defined modified-lateral technique of TLIP (mTLIP) block as a new approach. Ahiskalioglu et al. have reported that this approach has some advantages. Firstly, sonographic visualisation is more easily than the classical technique. Secondly, insertion of the needle from medial to lateral direction reduces the risk of possible neuraxial injection. It has been reported that this technique provides effective analgesia after lumbar spinal surgery.

The ultrasound (US) guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. at 2016 The ESPB contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves. ESPB provides thoracic analgesia at T5 level, abdominal analgesia at T7-9 level, and lumbar analgesia at T10-12, L3 level. In the literature, it has been reported that ESPB provides effective analgesia after lumbar spine surgery.

The aim of this study is to compare US-guided mTLIP block and ESPB for postoperative analgesia management after after lumbar disc herniation-laminectomy surgery. The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for lumbar disc herniation-laminectomy surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | The opioid consumption at perioperative period and postoperatively 24 hours
  The primary aim is to compare perioperative and postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Ahiskalioglu A, Alici HA, Selvitopi K, Yayik AM. Ultrasonography-guided modified thoracolumbar interfascial plane block: a new approach. Can J Anaesth. 2017 Jul;64(7):775-776. doi: 10.1007/s12630-017-0851-y. Epub 2017 Feb 27. No abstract available. PMID 28243853
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Ahiskalioglu A, Yayik AM, Doymus O, Selvitopi K, Ahiskalioglu EO, Calikoglu C, Alici HA, Karaca O. Efficacy of ultrasound-guided modified thoracolumbar interfascial plane block for postoperative analgesia after spinal surgery: a randomized-controlled trial. Can J Anaesth. 2018 May;65(5):603-604. doi: 10.1007/s12630-018-1051-0. Epub 2018 Jan 9. No abstract available. PMID 29318534